CLINICAL TRIAL: NCT06673537
Title: The Effects of Spinal Manipulation on Menstrual Symptoms, Pain Severity, and Sleep Quality in Individuals with Primary Dysmenorrhea
Brief Title: Spinal Manipulation for Menstrual Symptoms and Sleep in Individuals with Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Narges Piri (Other)
Collaborators: Rustem Mustafaoglu (Unknown)
Responsible Party: Sponsor-Investigator, Narges Piri, PT, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/208
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Primary Dysmenorrhea; Dysmenorrhea
Keywords: Connective Tissue Massage; CTM; Spinal Manipulation; SP; Physiotherapy; Massage; Menstrual Pain; Rehabilitation; Complementary Therapy; Women's Health; Manual Therapy; Pain Relief
MeSH Terms: conditions — Dysmenorrhea | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manip (Experimental): Manip: Connective Tissue Massage (CTM) + Spinal Manipulation (SM) Participants in the CTM+SM group will be applied three times a week, starting from the predicted day of ovulation (cycle length minus 14 days) until the onset of the next menstrual period. This will include treatment of the pelvic regions, specifically the sacral, lumbar, lower thoracic, and anterior pelvic areas. In addition to the CTM, spinal manipulation will be performed. The manipulation will follow the CTM and will involve the application of high-velocity, low-amplitude (HVLA) force bilaterally to all clinically relevant vertebral levels from T10 to L5, as well as to the sacroiliac joints, accompanied by an audible release from one or more joints. Treatment will be administered three times a week, with each session lasting 20 minutes. This regimen will continue for a duration of six weeks.
  Interventions: Other: Connective Tissue Massage (CTM); Other: Spinal Manipulation
- Sham Manip (Sham Comparator): Sham Manip: Connective Tissue Massage (CTM) + Sham Spinal Manipulation (Sham SM) The intervention will be applied three times a week, starting from the predicted day of ovulation (cycle length minus 14 days) until the onset of the next menstrual period. This will include treatment of the pelvic regions, specifically the sacral, lumbar, lower thoracic, and anterior pelvic areas. In addition to the CTM, sham spinal manipulation will be performed three times a week. This will involve the application of low-amplitude force bilaterally to all clinically relevant vertebral levels from T10 to L5 and to the sacroiliac joints, without producing any audible release. Treatment will be administered three times a week, with each session lasting 20 minutes. This regimen will continue for a duration of six weeks.
  Interventions: Other: Connective Tissue Massage (CTM); Other: Sham Spinal Manipulation
- Control Group (No Intervention): Participants in this group will undergo an initial assessment during which general information about the study will be provided. They will be informed about the importance of refraining from taking any medications throughout the six-week study period. All participants will be re-evaluated after the completion of the six weeks.

INTERVENTIONS:
Other: Connective Tissue Massage (CTM) — Connective Tissue Massage (CTM) was administered to the lumbar and abdominal regions by an experienced physiotherapist three times a week for 15 minutes over six weeks. The treatment started from the predicted day of ovulation (cycle length minus 14 days) until the onset of the next menstrual period. Both short and long strokes were utilized during CTM. Each stroke was repeated three times, first on the right side and then on the left side, across all manipulated areas. During the manipulation, the tip of the middle finger remained in contact with the patient's skin. The finger was positioned at a 45° angle, with the distal interphalangeal joint in flexion, and was moved to create traction.
  During the lumbar region treatment, participants were instructed to sit upright with their hips, knees, and ankles flexed at 90°, ensuring that their thighs and feet were fully supported. For the abdominal region treatment, participants lay supine with pillows placed under their head and knees.
  Arms: Manip; Sham Manip
Other: Spinal Manipulation — Spinal manipulation was performed by an experienced physiotherapist on the intervention group three times a week following Connective Tissue Massage (CTM). Participants in this group were positioned laterally, ensuring their lower leg remained straight and in contact with the treatment table. The contralateral or upper hip and knee were flexed and positioned so that they did not touch the table, allowing an unopposed force to be applied at the selected joint. Following CTM, manipulation was carried out with high-velocity, low-amplitude (HVLA) force applied bilaterally to all clinically relevant vertebral levels from T10 to L5 and the sacroiliac joints, accompanied by an audible sound from one or more joints.
  Arms: Manip
Other: Sham Spinal Manipulation — Sham spinal manipulation was administered by an experienced physiotherapist to the Sham Manipulation group three times a week following Connective Tissue Massage (CTM). In this group, participants were positioned laterally with their lower legs straight and in contact with the treatment table. The contralateral or upper hip and knee were flexed and positioned so that they did not touch the table, thereby allowing an unopposed force to be applied at the selected joint. Following CTM, low-amplitude force was applied bilaterally to all clinically relevant vertebral levels from T10 to L5 and the sacroiliac joints, without creating an audible sound.
  Arms: Sham Manip

SUMMARY:
The goal of this observational study is to evaluate if spinal manipulation (SM) combined with connective tissue massage (CTM) improves pain, menstrual symptoms, depression levels, and sleep quality in women with primary dysmenorrhea (PD). The main questions it aims to answer are:

Null Hypothesis (H0): SM has no effect on primary dysmenorrhea symptoms, pain severity, depression levels, or sleep quality.

Alternative Hypothesis (H1): SM has a significant effect on primary dysmenorrhea symptoms, pain severity, depression levels, and sleep quality.

Researchers will compare three groups to determine if the combined intervention improves menstrual health:

An intervention group receiving both KDM and SM applied to the abdominal and lumbar areas, A sham group receiving KDM with a sham SM procedure, A control group receiving no intervention.

Participants will:

Undergo three weekly sessions for one menstrual cycle (approximately three weeks), continuing for two cycles (six weeks total), Complete assessments on pain (VAS), menstrual symptoms (Menstrual Symptom Questionnaire), depression (Beck Depression Inventory), and sleep quality (Pittsburgh Sleep Quality Index) at the study's start and conclusion.

This study aims to provide new insights into the combined effects of KDM and SM on menstrual health, potentially guiding future rehabilitation interventions for PD.

DETAILED DESCRIPTION:
After experiencing primary dysmenorrhea, many individuals report significant menstrual symptoms, including pain severity and sleep disturbances, which can lead to decreased quality of life and increased dependence on medication for relief. In chronic cases, individuals with moderate to severe menstrual pain often exhibit functional deficits, impacting their daily living activities. This highlights the necessity for effective rehabilitation strategies that address both symptom management and overall quality of life.

Current treatment approaches for primary dysmenorrhea focus on pharmacological interventions, lifestyle modifications, and physiotherapy. The primary aim is to reduce pain severity and improve sleep quality through targeted therapies. Techniques such as spinal manipulation and connective tissue massage (KDM) have shown promise in promoting pain relief and enhancing functional outcomes. However, these techniques may not be universally applicable to all patients, particularly those with significant menstrual pain and associated sleep disturbances.

As outlined, promoting functional recovery in individuals with primary dysmenorrhea is crucial; however, the role of spinal manipulation and other manual therapies in this recovery process remains underexplored. Rehabilitation strategies must be tailored to individual needs and severity of symptoms. This study proposes a novel approach that integrates spinal manipulation with connective tissue massage, aimed at providing comprehensive relief and facilitating recovery in individuals with primary dysmenorrhea.

The proposed intervention includes both spinal manipulation and KDM, administered by trained physiotherapists. This dual approach is designed to address pain at its source and improve overall musculoskeletal function. Evidence suggests that combined therapies may lead to enhanced neurophysiological responses, promoting both pain relief and functional improvements.

The underlying mechanisms of action for this combined approach may involve multiple pathways. Spinal manipulation may facilitate increased blood flow and reduce muscle tension, while KDM is thought to enhance tissue pliability and alleviate discomfort. Together, these interventions may induce neuroplastic changes, facilitating improved pain management and functional outcomes.

To date, studies on combined therapeutic approaches for primary dysmenorrhea have demonstrated promising results, including reduced pain severity and improved sleep quality. However, research specifically focusing on the synergistic effects of spinal manipulation and KDM remains limited. This study aims to evaluate the efficacy of this integrated approach on menstrual symptoms, pain severity, and sleep quality in individuals suffering from primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Having primary dysmenorrhea according to the criteria specified in the Primary Dysmenorrhea Consensus Guide (1. Onset of pain 6 to 24 months after menarche, 2. Pain lasting between 8 to 72 hours, and 3. The most intense pain occurring on the 1st and/or 2nd day of menstruation),
* Having a regular menstrual cycle (28 ± 7 days).

Exclusion Criteria:

* Having gastrointestinal, urogenital, autoimmune, or psychiatric disorders (serious psychiatric disorders that would prevent participation in the study),
* Having other chronic pain syndromes,
* Having given birth or a positive pregnancy test,
* Using an intrauterine device (IUD),
* Having undergone pelvic surgery,
* Having used chronic medications, including oral contraceptives or antidepressants, within at least 6 months prior to the study,
* Having irregular menstrual cycles (shorter than 21 days or longer than 35 days, and/or a cycle variation exceeding 4 days),
* Having a history of pathological conditions indicating secondary dysmenorrhea.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only self-identified females are eligible to participate in this study, as it specifically addresses menstrual-related issues.
Enrollment: 75 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-09-16 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, post-intervention (approximately 6 weeks)
  The Visual Analog Scale (VAS) is a subjective measure used to assess the intensity of participants' pain. Participants are asked to indicate their perceived level of pain on a 10 cm line. One end of the line is marked as 0, indicating no pain, while the other end is marked as 10, representing unbearable pain.
  Participants were instructed to mark the intensity of pain experienced during the first three days of their initial menstrual period before joining the study, as well as during the last menstrual period at the end of the study, on three separate VAS lines, with the highest value recorded. The VAS is considered a valid and reliable tool for measuring experimental and clinical pain, demonstrating high sensitivity in detecting changes in clinical pain treatment and small variations in pain intensity.
Menstrual Symptom Questionnaire (MSQ) | Baseline, post-intervention (approximately 6 weeks)
  The Menstrual Symptom Questionnaire (MSQ) is a 22-item five-point Likert-type questionnaire developed by Chesney and Tasto (1975) to assess menstrual pain and symptoms. In 2014, Güvenç and colleagues adapted this questionnaire into Turkish, ensuring its validity. The questionnaire consists of three subscales: menstrual pain symptoms, negative effects/somatic complaints, and coping strategies. The questionnaire is scored between 22 and 110, with an increase in the average score indicating a greater severity of menstrual symptoms. The questionnaire was administered face-to-face to participants before and after the study, and their responses were recorded.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, post-intervention (approximately 6 weeks)
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire developed to assess sleep quality and disturbances over a one-month period. It consists of 19 self-rated questions and 5 questions rated by a bed partner or roommate. The PSQI was adapted into Turkish in 2014 by Güvenç and colleagues, ensuring its validity. The questionnaire evaluates seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores range from 0 to 21, with higher scores indicating worse sleep quality. The questionnaire was administered face-to-face to participants before and after the study, and their responses were recorded.
Beck Depression Inventory (BDI) | Baseline, post-intervention (approximately 6 weeks)
  The Beck Depression Inventory (BDI) was used to assess the risk of depression and determine the level of depressive symptoms, with its Turkish validity and reliability established by Hisli. The inventory consists of 21 categories, each with four options. Each item is scored between 0 and 3, resulting in a total score ranging from 0 to 63. Scores are categorized as follows: 0-9 = Minimal depressive symptoms, 10-16 = Mild depressive symptoms, 17-29 = Moderate depressive symptoms, and 30-63 = Severe depressive symptoms. The questionnaire was administered face-to-face to participants before and after the study, and their responses were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Narges PIRI, Bcs, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Graduate Studies, Department of Physiotherapy and Rehabilitation; Rüstem MUSTAFAOĞLU PT, PhD, Study Chair — Istanbul University-Cerrahpasa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul, Istanbul
  - IstanbulUC, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) due to confidentiality concerns and the need to protect participant privacy. Additionally, our study is designed to aggregate data for analysis, focusing on group outcomes rather than individual results. This approach aligns with our ethical obligations and the guidelines set forth by our institution.

REFERENCES:
- [Background] Hernandez-Diaz S, Garcia-Rodriguez LA. Epidemiologic assessment of the safety of conventional nonsteroidal anti-inflammatory drugs. Am J Med. 2001 Feb 19;110 Suppl 3A:20S-7S. doi: 10.1016/s0002-9343(00)00682-3. PMID 11173046
- [Background] Hailemeskel S, Demissie A, Assefa N. Primary dysmenorrhea magnitude, associated risk factors, and its effect on academic performance: evidence from female university students in Ethiopia. Int J Womens Health. 2016 Sep 19;8:489-496. doi: 10.2147/IJWH.S112768. eCollection 2016. PMID 27695366
- [Background] Eryilmaz G, Ozdemir F, Pasinlioglu T. Dysmenorrhea prevalence among adolescents in eastern Turkey: its effects on school performance and relationships with family and friends. J Pediatr Adolesc Gynecol. 2010 Oct;23(5):267-72. doi: 10.1016/j.jpag.2010.02.009. Epub 2010 May 21. PMID 20493741
- [Background] Molins-Cubero S, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, Heredia-Rizo AM, Bosca-Gandia JJ, Ricard F. Changes in pain perception after pelvis manipulation in women with primary dysmenorrhea: a randomized controlled trial. Pain Med. 2014 Sep;15(9):1455-63. doi: 10.1111/pme.12404. Epub 2014 Mar 25. PMID 24666560
- [Background] Ozgul S, Uzelpasaci E, Orhan C, Baran E, Beksac MS, Akbayrak T. Short-term effects of connective tissue manipulation in women with primary dysmenorrhea: A randomized controlled trial. Complement Ther Clin Pract. 2018 Nov;33:1-6. doi: 10.1016/j.ctcp.2018.07.007. Epub 2018 Jul 21. PMID 30396605
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671